CLINICAL TRIAL: NCT04544072
Title: A Prospective Analysis of the Quality and Quantity of Antibiotic Prescriptions for Bacterial Respiratory Tract Superinfection in Patients Hospitalized in COVID-19 Wards of a Tertiary University Hospital During the COVID-19 Pandemic
Brief Title: Analysis of the Quality and Quantity of Antibiotic Prescriptions for Bacterial Respiratory Tract Superinfection in Patients Hospitalized in COVID-19 Wards
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Johan Van Laethem, Principal investigator, Universitair Ziekenhuis Brussel
Other Study IDs: 2020-163
Record Dates: First submitted 2020-08-15; First posted 2020-09-10 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: SARS-CoV Infection; Antimicrobial Stewardship; Respiratory Tract Infections; Antibiotic Resistance
Keywords: respiratory tract infection; antimicrobial stewardship; SARS-CoV infection; COVID-19; Antibiotic resistance
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; Respiratory Tract Infections; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this prospective observational study, a quantitative and qualitative analysis of antibiotic prescriptions for presumed respiratory tract (super)infection in patients hospitalized on COVID-19 wards will be made.

Drivers of antibiotic prescription for presumed respiratory tract infection in patients suspected of being infected with COVID-19 or with definite COVID-19 infections will be identified.

DETAILED DESCRIPTION:
Patients hospitalized on a COVID-19 ward for more than 24 hours will be included. Those with one or more antimicrobial prescription(s) for a presumed respiratory tract (super)infection will be identified and every antibiotic dose will be scored as appropriate, inappropriate, suboptimal or unnecessary by at least two infectious disease (ID) specialists, on an independent manner. If the scoring of the two ID specialists will defer, a third ID specialist will come to a conclusion after discussion with the two other ID specialists.

A quantification of the total amount of antibiotics, prescribed for presumed respiratory tract (super)infection will be made for patients with a COVID-19 diagnosis, but also a quantification for every category of appropriateness will be made.

Possible drivers like the degree of hypoxemia, laboratory parameters, qSOFA score, duration of symptoms, age, comorbidities, symptoms,... associated with the prescription of antimicrobials for a presumed respiratory tract (sur)infection will be identified.

ELIGIBILITY:
Inclusion Criteria:

* Men and women hospitalized in one of the COVID wards (no data will be collected during a stay on the ICU department) of UZ Brussel for more than 24 hours and willing to sign the informed consent form (or signed by one of their legal representative(s) if unable).

Exclusion Criteria:

* patients younger than 18 years old
* patients not willing to sign the informed consent form
* patients hospitalized for a shorter duration than 24 hours on a COVID-19 ward

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients fulfilling the above mentioned inclusion criteria, hospitalized on a COVID-19 ward, having signed the informed consent form (ICF) by themselves or by one of their legal representatives.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
Total antimicrobial consumption for suspicion of secondary bacterial respiratory infections in hospitalized patients in COVID wards with a clinical or PCR-based COVID diagnosis, expressed as 'Daily defined doses/hospitalization'. | 7 months
  The total antibiotic use, expressed as Daily Defined Doses (DDD) of antibiotics in grams. This will be aggregated with the amount of hospitalizations to arrive at one reported value: DDD/hospitalization (expressed as grams/hospitalization), for every antibiotic and antibiotic formulation (IV or PO) separately but also for all prescribed antibiotics in general.
Total antimicrobial consumption for suspicion of secondary bacterial respiratory infections in hospitalized patients in COVID wards with a clinical or PCR-based COVID diagnosis, expressed as 'Daily defined doses/1000 hospitalized patient days'. | 7 months
  The total antibiotic use, expressed as Daily Defined Doses (DDD) in grams. This will be aggregated with the total amount of hospitalized patient days to arrive at one reported value: DDD/1000 hospitalization patient days (expressed as grams/1000 hospitalization days), for every antibiotic and antibiotic formulation (IV or PO) separately but also for all prescribed antibiotics in general. 1000 hospitalised patient days for every antibiotic and antibiotic formulation (IV or PO) separately but also for all prescribed antibiotics in general.
Total antimicrobial consumption for suspicion of secondary bacterial respiratory infections in hospitalized patients in COVID wards with a clinical or PCR-based COVID diagnosis, expressed as 'Daily doses of administration/hospitalization'. | 7 months
  The total antibiotic use, expressed as Daily Doses of Administration (DDA) of antibiotics in grams. This will be aggregated with the amount of hospitalizations to arrive at one reported value: DDA/hospitalization (expressed as grams/hospitalization), for every antibiotic and antibiotic formulation (IV or PO) separately but also for all prescribed antibiotics in general.
Total antimicrobial consumption for suspicion of secondary bacterial respiratory infections in hospitalized patients in COVID wards, expressed as 'Daily doses of administration (DDA)/1000 hospitalized patient days'. | 7 months
  The total antibiotic use, expressed as Daily Doses of Administration (DDA) in grams. This will be aggregated with the total amount of hospitalized patient days to arrive at one reported value: DDA/1000 hospitalization patient days (expressed as grams/1000 hospitalization days), for every antibiotic and antibiotic formulation (IV or PO) separately but also for all prescribed antibiotics in general.

SECONDARY OUTCOMES:
The degree of appropriateness of antimicrobial prescriptions for presumed respiratory tract (super)infection | 7 months
  The degree of appropriateness for each antibiotic (AB) formulation separately but also for all prescribed antibiotics in general, with distinction between 'Appropriate', 'Unnecessary', 'inappropriate' and 'suboptimal' AB choice. Results will be expressed as DDD or DDA of appropriate AB/1000 patient days, DDD or DDA of unnecessary AB/1000 patient days, DDD or DDA of inappropriate AB/1000 patient days and DDD or DDA of suboptimal AB/1000 patient days. Used units: g/1000 hospitalized patients days
The degree of appropriateness of antimicrobial prescriptions for presumed respiratory tract (super)infection, denominator 2 | 7 months
  The degree of appropriateness for each antibiotic (AB) formulation separately but also for all prescribed antibiotics in general, with distinction between 'Appropriate', 'Unnecessary', 'inappropriate' and 'suboptimal' AB choice. Results will be expressed as DDD or DDA of appropriate AB/hospitalization, DDD or DDA of unnecessary AB/hospitalization, DDD or DDA of inappropriate AB/hospitalization and DDD or DDA of suboptimal AB/hospitalization. Used units: g/hospitalization
Rate of Clostridioides Difficile infections | 7 months
  The number of C. Difficile infections in the inpatient setting
Is there a significant difference in age comparing the group receiving antibiotics for a suspicion of COVID-19 superinfection and the group without antibiotics? | 7 months
  median or mean age (number) , comparing the group receiving antibiotics for a suspicion of COVID-19 superinfection and the group without antibiotics?
Is there a significant difference in weight comparing the group receiving antibiotics for a suspicion of COVID-19 superinfection and the group without antibiotics? | 7 months
  median or mean weight (kg), comparing the group receiving antibiotics for a suspicion of COVID-19 superinfection and the group without antibiotics?
significant difference in amount of comorbidities comparing the group receiving antibiotics for a suspicion of COVID-19 superinfection and the group without antibiotics? | 7 months
  rate of comorbidities expressed as mean Charlson Comorbidity Index score, comparing the group receiving antibiotics for a suspicion of COVID-19 superinfection and the group without antibiotics
significant difference in rate of chronical pulmonary disease as a comorbidity, comparing the group receiving antibiotics for a suspicion of COVID-19 superinfection and the group without antibiotics? | 7 months
  rate of chronical pulmonary disease, comparing the group receiving antibiotics for a suspicion of COVID-19 superinfection and the group without antibiotics
significant difference in rate of haematological or solid neoplasia as a comorbidity, comparing the group receiving antibiotics for a suspicion of COVID-19 superinfection and the group without antibiotics? | 7 months
  rate of haematological or solid neoplasia, comparing the group receiving antibiotics for a suspicion of COVID-19 superinfection and the group without antibiotics
significant difference in rate of diabetes mellitus as a comorbidity, comparing the group receiving antibiotics for a suspicion of COVID-19 superinfection and the group without antibiotics? | 7 months
  rate of diabetes mellitus, comparing the group receiving antibiotics for a suspicion of COVID-19 superinfection and the group without antibiotics
significant difference in rate of patients with presence or not of at least one suggestive symptom of COVID-19 symptomatology, comparing the group receiving antibiotics for a suspicion of COVID-19 superinfection and the group without antibiotics? | 7 months
  rate of patients with fever (t°>38°c), dyspnea, cough, runny nose, throat pain, thoracic pain, myalgia, fatigue, anosmia, confusion at admission, comparing the group receiving antibiotics for a suspicion of COVID-19 superinfection and the group without antibiotics?
significant difference in rate of patients with recent AB prescription, comparing the group receiving antibiotics for a suspicion of COVID-19 superinfection and the group without antibiotics? | 7 months
  rate of patients rate of patients having received an antibiotic prescription for a suspicion of respiratory tract infection during the 3 weeks before hospitalization, comparing the group receiving antibiotics for a suspicion of COVID-19 surinfection and the group without antibiotics?
Is there a significant difference in the rate of patients having had at least one positive significant respiratory germ culture, comparing the group receiving antibiotics for a suspicion of COVID-19 superinfection and the group without antibiotics? | 7 months
  rate of patients with significant positive respiratory cultures, comparing the group receiving antibiotics for a suspicion of COVID-19 superinfection and the group without antibiotics?
Is there a significant difference in the rate of patients needing oxygen supletion at day 1 of hospitalization, comparing the group receiving antibiotics for a suspicion of COVID-19 superinfection and the group without antibiotics? | 7 months
  rate of patients with oxygen suppletion need, comparing the group receiving antibiotics for a suspicion of COVID-19 superinfection and the group without antibiotics?
significant difference in the mean duration of hospitalization, comparing the group receiving antibiotics for a suspicion of COVID-19 superinfection and the group without antibiotics? | 7 months
  mean duration of hospitalization on a COVID-ward, comparing the group receiving antibiotics for a suspicion of COVID-19 superinfection and the group without antibiotics?
significant difference in the rate of ICU admission, comparing the group receiving antibiotics for a suspicion of COVID-19 superinfection and the group without antibiotics? | 7 months
  rate of ICU admission, comparing the group receiving antibiotics for a suspicion of COVID-19 superinfection and the group without antibiotics?
Is there a significant difference in the mean value of oxygen saturation percentage over fractional oxygen percentage, comparing the group receiving antibiotics for a suspicion of COVID-19 superinfection and the group without antibiotics? | 7 months
  mean SatO2/FiO2 ratio (number ranging from 50-500), comparing the group receiving antibiotics for a suspicion of COVID-19 superinfection and the group without antibiotics?
Is there a significant difference in qSOFA score level at admission, comparing the group receiving antibiotics for a suspicion of COVID-19 superinfection and the group without antibiotics? | 7 months
  mean/median qSOFA score at admission, comparing the group receiving antibiotics for a suspicion of COVID-19 superinfection and the group without antibiotics?
Is there a significant difference in the rate of lymphopenia, comparing the group receiving antibiotics for a suspicion of COVID-19 superinfection and the group without antibiotics? | 7 months
  Rate of lymphopenia (<1250/mcl), comparing the group receiving antibiotics for a suspicion of COVID-19 superinfection and the group without antibiotics?
significant difference in the mean value of C-reactive protein measured at day 1 of hospitalization on a COVID-ward ,comparing the group receiving antibiotics for a suspicion of COVID-19 superinfection and the group without antibiotics? | 7 months
  mean CRP values (mg/dl) at day 1 of hospitalization, comparing the group receiving antibiotics for a suspicion of COVID-19 superinfection and the group without antibiotics
significant difference in the mean value of white blood cell count measured at day 1 of hospitalization on a COVID-ward ,comparing the group receiving antibiotics for a suspicion of COVID-19 superinfection and the group without antibiotics? | 7 months
  mean WBC count (/mcl) values at day 1 of hospitalization, comparing the group receiving antibiotics for a suspicion of COVID-19 superinfection and the group without antibiotics
significant difference in the mean value of neutrophil count measured at day 1 of hospitalization on a COVID-ward ,comparing the group receiving antibiotics for a suspicion of COVID-19 superinfection and the group without antibiotics? | 7 months
  mean neutrophil count (/mcl) values at day 1 of hospitalization, comparing the group receiving antibiotics for a suspicion of COVID-19 superinfection and the group without antibiotics
significant difference in the mean value of lymphocyte count measured at day 1 of hospitalization on a COVID-ward ,comparing the group receiving antibiotics for a suspicion of COVID-19 superinfection and the group without antibiotics? | 7 months
  mean lymphocyte count (/mcl) values at day 1 of hospitalization, comparing the group receiving antibiotics for a suspicion of COVID-19 surinfection and the group without antibiotics
significant difference in the mean value of creatinine measured at day 1 of hospitalization on a COVID-ward ,comparing the group receiving antibiotics for a suspicion of COVID-19 superinfection and the group without antibiotics? | 7 months
  mean creatinine (mg/dl) values at day 1 of hospitalization, comparing the group receiving antibiotics for a suspicion of COVID-19 superinfection and the group without antibiotics
significant difference in the mean value of LDH measured at day 1 of hospitalization on a COVID-ward ,comparing the group receiving antibiotics for a suspicion of COVID-19 superinfection and the group without antibiotics? | 7 months
  mean LDH (U/L) values at day 1 of hospitalization, comparing the group receiving antibiotics for a suspicion of COVID-19 superinfection and the group without antibiotics
significant difference in the mean value of bilirubin measured at day 1 of hospitalization on a COVID-ward ,comparing the group receiving antibiotics for a suspicion of COVID-19 superinfection and the group without antibiotics? | 7 months
  mean bilirubin (mg/dl) values at day 1 of hospitalization, comparing the group receiving antibiotics for a suspicion of COVID-19 superinfection and the group without antibiotics
significant difference in the mean value of ferritin (first value during hospitalization),comparing the group receiving antibiotics for a suspicion of COVID-19 superinfection and the group without antibiotics? | 7 months
  mean ferritin (mcg/l) values, comparing the group receiving antibiotics for a suspicion of COVID-19 superinfection and the group without antibiotics
significant difference in the mean value of troponins (first value during hospitalization),comparing the group receiving antibiotics for a suspicion of COVID-19 superinfection and the group without antibiotics? | 7 months
  mean troponin (mcg/l) values, comparing the group receiving antibiotics for a suspicion of COVID-19 superinfection and the group without antibiotics
significant difference in the mean value of D-dimers (first value during hospitalization),comparing the group receiving antibiotics for a suspicion of COVID-19 superinfection and the group without antibiotics? | 7 months
  mean D-dimer (ng/ml) values, comparing the group receiving antibiotics for a suspicion of COVID-19 superinfection and the group without antibiotics

CONTACTS AND LOCATIONS:
Overall Officials: Johan Dr Van Laethem, MD, Principal Investigator — Principal Investigator
Locations (1):
- UZ Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Van Laethem J, Wuyts S, Van Laere S, Dirkx S, Seyler L, Mertens R, Ilsen B, Lacor P, Pierard D, Allard SD. Antibiotic Prescriptions Targeting Bacterial Respiratory Infections in Admitted Patients with COVID-19: A Prospective Observational Study. Infect Dis Ther. 2021 Dec;10(4):2575-2591. doi: 10.1007/s40121-021-00535-2. Epub 2021 Sep 16. PMID 34529255